CLINICAL TRIAL: NCT01197976
Title: Double-blind, Randomized, Right-left Study Comparing TEPSO® Socks With Standard Socks in Improving Palmoplantar Psoriasis
Brief Title: Efficacy Study of TEPSO® Socks in Improving Palmoplantar Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lenzi Egisto S.P.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEPSO1
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Palmoplantar Psoriasis
Keywords: psoriasis; soles; teflon
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEPSO socks (Experimental): This arm include all patients sides (left or right) treated with TEPSO socks.
  Interventions: Device: TEPSO cloth
- Standard socks (Placebo Comparator): This arm include all patients sides (left or right) treated with standard cotton socks.
  Interventions: Device: Standard cloth

INTERVENTIONS:
Device: TEPSO cloth — TEPSO stocks should be worn continuously for 4 weeks of the study and will be changed every 3 days without wearing again those already used (even after washing).
  Other Names: Teflon
  Arms: TEPSO socks
Device: Standard cloth — Standard cotton stocks should be worn continuously for 4 weeks of the study and will be changed every 3 days without wearing again those already used (even after washing).
  Other Names: cotton
  Arms: Standard socks

SUMMARY:
The purpose of this study is to evaluate the efficacy of a special sock, manufactured using TEPSO®, compared to a normal cotton sock in the prognosis of symmetrical palmoplantar psoriasis present for at least one year.

DETAILED DESCRIPTION:
The clinical manifestations of palmoplantar psoriasis have an important impact on well being and quality of life. The manifestation of the disease is often exacerbated by factors such as significant physical and mechanical stress resulting from repeated and prolonged pressure over the affected areas and by everyday clothing. These problems have led the textile industry Lenzi Egisto S.p.A. to conduct some preliminary analyses to find a fabric that meets the specific needs of psoriatic patients in relation to everyday clothing. This preliminary study led to the creation of a particular fabric, TEPSO®, with features specific to the identified needs. This material consists essentially of PTFE (commercially known as Teflon®) and thus presents interesting characteristics that make it suitable for creating garments for patients with psoriasis:

* Excellent flow properties and low surface friction
* non-stick
* Complete biocompatibility and chemical inertness

We can therefore speculate that in palmoplantar psoriasis high smoothness of the fabric and low coefficient of friction may translate into less discomfort felt by patients during normal physical activities, and into improved clinical course of the disease. In the end, it is expected that reduced mechanical compression and friction, would result into partial or complete clinical remission within a few weeks of use.

Therefore we propose to conduct a randomized controlled, double-blind, left-right clinical trial to assess the hypothesis that in palmoplantar psoriasis the use of TEPSO® could induce an improvement of disease and overall quality of life. To better assess the effects of treatment, the use of clothing in the study will be limited to symmetrical psoriatic lesions of feets in order to include areas that are comparable and relevant from a functional point of view.

ELIGIBILITY:
Inclusion Criteria:

* Palmoplantar psoriasis present for at least one year
* Symmetrical foot lesions with at least 5% of the skin surface involvement
* Difference less than or equal to 10% extension of lesions on both sides of the body
* Suspension for over 3 months from start of the study of any systemic drugs for psoriasis, immunosuppressive treatments (cyclosporine, systemic steroids), psoralen plus ultraviolet A irradiation (PUVA) or ultraviolet B phototherapy (UVB)

Exclusion Criteria:

* Nonsymmetrical foot lesions or less than 5% of the skin surface involvement
* Difference of more than 10% extension of lesions on both sides of the body
* Patients who have performed, within 3 months before inclusion in the study, treatments with systemic drugs for psoriasis, immunosuppressive treatments (cyclosporine, systemic steroids), psoralen plus ultraviolet A irradiation (PUVA) or ultraviolet B phototherapy (UVB)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percentage reduction of treated areas from baseline | 4 weeks
  Percentage reduction is based on standardized photos and computerized image evaluation

SECONDARY OUTCOMES:
Quality of life | 4 weeks
  Quality of life is assessed by patient with visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Naldi, dermatology, Study Director — Centro Studi Gised
Locations (3):
- Italy (3):
  - Department of Dermatology, "Tor Vergata" general hospital, Rome, Lazio
  - Department of Dermatology, Fondazione S.Raffaele del monte Tabor, Milan, Lombardy
  - Department of Dermatology, USL 4, Prato, Tuscany